CLINICAL TRIAL: NCT06777420
Title: Question Prompt List as a Tool to Promote Patient-physician Concordance in the Understanding of Information on Neoadjuvant Treatment in Breast Cancer: a Randomized Controlled Trial
Brief Title: Question Prompt List in Breast Cancer Patients Planned for Neoadjuvant Chemotherapy
Acronym: QPL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 280103
Record Dates: First submitted 2025-01-03; First posted 2025-01-15 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); Neoadjuvant Therapy; Shared Decision Making
Keywords: breast cancer; neoadjuvant therapy; question prompt list; patient-physician communication; shared decision making
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Question prompt list (Experimental): Patients will receive a question prompt list before their 1st visit to the oncologist for discussion about neoadjuvant therapy
  Interventions: Other: Question prompt list
- Usual care (No Intervention): Patients do not receive a question prompt list before their 1st visit to the oncologist

INTERVENTIONS:
Other: Question prompt list — The question prompt list includes 12 questions related to neoadjuvant therapy. It has been developed by an expert team including breast surgeons, oncologists, nurses, and psychologists and has been refined through focus interview with patient advocates and caregivers.
  Arms: Question prompt list

SUMMARY:
Preoperative chemotherapy has been shown to be at least as effective as postoperative chemotherapy in breast cancer patients and has seen increased use over time. The decision regarding neoadjuvant treatment is complex, as various aspects need to be considered, and the patient's role in the decision-making process is central.

The information provided by doctors to patients about preoperative treatment can be complicated, including details about treatment options, treatment plans, and side effects. If this information is not conveyed adequately, there is a risk of misunderstandings, which can lead to increased anxiety and stress for patients regarding their decisions.

In oncology, question prompt lists (QPL) have been used as a tool to support patients by improving the information conveyed by doctors in various contexts where complex decisions need to be made. Studies have shown that QPL can facilitate better information exchange. However, their use in discussions about preoperative treatment for breast cancer patients has not been studied. Furthermore, evidence from randomized studies on the use of QPL in clinical practice is very limited.

The aim of this study is to investigate whether the use of QPL during patient consultations involving discussions about neoadjuvant chemotherapy can improve information exchange in various aspects: understanding of the treatment; anxiety about the decision; participation in the decision-making process; patient-doctor communication; and decision-related conflict.

ELIGIBILITY:
Inclusion Criteria:

* Patients with operable breast cancer eligible for systemic neoadjuvant therapy, according to current treatment guidelines.

Exclusion Criteria:

* Patients with locally advanced breast cancer where neoadjuvant therapy is mandatory rather than a treatment option.
* Patients with cognitive impairment that are assessed from treating physician as unable to participate.
* Patients who cannot speak/read neither Swedish nor English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Concordance rate between patient and oncologist | Within five days from patient visit
  Concordance rate regarding the information that was given from oncologist to the patient during the patient visit.

SECONDARY OUTCOMES:
Level of anxiety | Within five days from patient visit
  The level of anxiety (measured by the State-Trait Anxiety Inventory) after patient visit to oncologist and before treatment initiation.
Decision-making participation | Within five days from patient visit
  Patients' perception about their participation in decision-making process (measured by the 9-item Shared Decision Making Questionnaire)
Patient-physician communication | Within five days from patient visit
  Patients' experience on patient-physician communication (measured by the Patient Satisfaction Questionnaire and the Perceived Efficacy in Patient-Physician Interactions)
Decisional conflict | Within five days from patient visit
  Patients' experience on decisional conflict (measured by the decisional conflict scale)

CONTACTS AND LOCATIONS:
Overall Officials: Antonis Valachis, MD, PhD, Principal Investigator — Department of Oncology, Örebro University Hospital, Sweden
Locations (3):
- Sweden (3):
  - Akademiska Uppsala University Hospital, Uppsala, Region Uppsala
  - Västerås General Hospital, Västerås, Region Västmanland
  - Örebro University Hospital, Örebro